CLINICAL TRIAL: NCT02057887
Title: Safety,Tolerability and Pharmacokinetic Study of Recombinant Human Interferon Alfa 2B in Chronic Hepatitis C Patients (HM10660A)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-IFN-201
Record Dates: First submitted 2013-08-08; First posted 2014-02-07 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Chronic Hepatitis C Virus Genotype I
MeSH Terms: interventions — peginterferon alfa-2a

ARMS (4):
- Cohort1 (Experimental): HM10660A SC once weekly
  Interventions: Drug: HM10660A
- Cohort2 (Experimental): HM10660A SC once every 2 weeks
  Interventions: Drug: HM10660A
- Cohort3 (Experimental): HM10660A SC once every 4 weeks
  Interventions: Drug: HM10660A
- Cohort4 (Active Comparator): 180 mcg Pegasys SC once weekly
  Interventions: Drug: Pegasys

INTERVENTIONS:
Drug: HM10660A
  Other Names: Laps-IFNa
  Arms: Cohort1; Cohort2; Cohort3
Drug: Pegasys — 180 mcg Pegasys SC once weekly
  Arms: Cohort4

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of multiple ascending doses of HM10660A in subjects with chronic hepatitis C(HCV).

DETAILED DESCRIPTION:
* To evaluate the repeat-dose pharmacokinetics (PK) of HM10660A when given by weekly, biweekly, and monthly subcutaneous (SC) injection.
* To evaluate the repeat-dose pharmacodynamics (PD) of HM10660A when given by weekly, biweekly, and monthly SC injection.
* To explore the antiviral activity of HM10660A at Week 4, Week 12, and Week 24.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 65 years old, inclusive
* Willing and able to provide written informed consent.
* Previously untreated HCV infection with HCV RNA > 75,000 IU/mL at screening.
* HCV genotype 1a or 1b.
* Body mass index (BMI) between 18 and 38 kg/m2.
* Willing and able to comply with the protocol and available to complete the study schedule of assessments.

Exclusion Criteria:

* Pregnant women or women who may wish to become pregnant during the course of the study.
* Males and females of reproductive potential who are unwilling to use 2 forms of effective birth control throughout the duration of study treatment and for at least 6 months after the last dose of RBV. One method should include a condom with spermicide for males. Males must agree to refrain from sperm donation for at least 6 months after the last dose of RBV.
* Evidence of infection or co-infection with a non-genotype 1 HCV strain.
* Co-infection with hepatitis B virus (HBV) or human immunodeficiency virus (HIV).
* Lactating females

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
HCV RNA Viral load | Through study week 32
Safety/tolerability | Through study week 32
  symptom-directed physical examination, Vital signs, Inspection of the Injection site, Complete Physical examination, 12-lead ECG, Hematology/coagulation

SECONDARY OUTCOMES:
Rapid virologic response (RVR) | Study Week 4
Early virologic response (EVR) | Study week 12
Sustained virologic response (SVR) | Study week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Hanmi Clinical, Estado de México, State of Mexico, Mexico